CLINICAL TRIAL: NCT04446962
Title: LOC-R01: Randomized Phase IB/II Study of Escalating Doses of Lenalidomide and Ibrutinib in Association With R-MPV as a Targeted Induction Treatment for Patients Aged 18 to 60 (up to 65 for Phase II) With a Newly Diagnosed Primary Central Nervous System Lymphoma
Brief Title: LOC-R01 Study of Lenalidomide and Ibrutinib in Association With Rituximab-Methotrexate Procarbazine Vincristin (R-MPV)
Acronym: LOC-R01
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institut Curie (Other)
Collaborators: National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IC 2019-02; 2019-003632-23 (EudraCT Number)
Record Dates: First submitted 2020-06-22; First posted 2020-06-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Lymphoma, Large B-Cell, Diffuse; Central Nervous System Neoplasms, Primary
Keywords: Lymphoma; Nervous System; Primary
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Central Nervous System Neoplasms; Lymphoma; Neurologic Manifestations | interventions — Lenalidomide; ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: R-MPV with Lenalidomide (Active Comparator): Lenalidomide in association with R-MPV as a targeted induction treatment
  Interventions: Drug: Lenalidomide
- Arm B: R-MPV with Ibrutinib (Active Comparator): Ibrutinib in association with R-MPV as a targeted induction treatment
  Interventions: Drug: Ibrutinib

INTERVENTIONS:
Drug: Lenalidomide — Patients will receive 4 cycles of induction chemotherapy with R-MPV + Lenalidomide using the Maximum Tolerated Dose (MTD) of Lenalidomide and Ibrutinib as determined in the phase-Ib part of the study.
  Other Names: Revlimid
  Arms: Arm A: R-MPV with Lenalidomide
Drug: Ibrutinib — Patients will receive 4 cycles of induction chemotherapy with R-MPV + Ibrutinib, using the Maximum Tolerated Dose (MTD) of Lenalidomide and Ibrutinib as determined in the phase-Ib part of the study.
  Other Names: Imbruvica
  Arms: Arm B: R-MPV with Ibrutinib

SUMMARY:
This study is to improve the first-line induction chemotherapy, by combining either Ibrutinib, or Lenalidomide, to a conventional immuno- chemotherapy of R-MPV type (Rituximab-Methotrexate-Procarbazine-Vincristine). This is a randomized Phase II trial, preceded by a dose escalation phase Ib. The objective of the phase Ib is to rule out any limiting toxicity of the new treatment associations, and to determine the recommended dose of Lenalidomide and Ibrutinib to be used in the phase II. In the phase II study, patients will receive 4 cycles of R-MPV + Lenalidomide or 4 cycles of R-MPV + Ibrutinib. The therapeutic response will be evaluated after the 2nd and the 4th cycle. Patients in good therapeutic response will proceed to the consolidation phase with Autologous Stem Cell Transplantation (ASCT).

DETAILED DESCRIPTION:
The objective of this proposal is to test the feasibility and efficacy of two targeted induction chemotherapies obtained by adding either Lenalidomide or Ibrutinib to a standard Rituximab-High Dose (HD) Methotrexate (MTX) based induction chemotherapy regimen. The R-MPV regimen is chosen as the backbone chemotherapy because of its wide use with robust reproducible results and a good and manageable toxicity profile

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed Primary Central Nervous System Lymphoma (PCNSL).
2. a) Aged between 18 and 60 (>18 and < 60) - phase IB b) Aged between 18 and 65 (≥ 18 and ≤ 65) - phase II.
3. Histological confirmed diagnosis of Primary central nervous system lymphoma of Diffuse Large B-Cell Lymphomas (DLBCL) type OR patients with a measurable typical cerebral lesion on MRI with a diagnosis made by cytology and/or by flow cytometry on the vitreous or on the cerebral spinal fluid.
4. Measurable lesion on MRI with gadolinium enhancement.
5. Adequate hematological, renal and hepatic function (Laboratory Parameters realized within 14 days before inclusion):

   1. Absolute neutrophil count (ANC) >1000/mm3
   2. Platelets > 100,000/mm3 independent of transfusion support
   3. Alanine aminotransferase and aspartate aminotransferase ≤ 3 x Upper Limit of Normal (ULN)
   4. Total bilirubin ≤ 1.5 x ULN unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin
   5. Estimated Glomerular Filtration Rate ≥ 60 mL/min/1.73m2.
6. Able to swallow capsules.
7. Karnofsky performance status: 40-100% for the phase IB and no restriction on the KPS for the phase II.
8. Able to understand teratogenic risks of the Lenalidomide and Ibrutinib. Patient must be able to understand and fulfill the Lenalidomide Pregnancy Prevention Plan requirements. This plan may be accepted by the person of confidence in case of impaired cognitive status of the patient.
9. Women of childbearing potential (WCBP)* and men who are sexually active must be practicing a highly effective method** of birth control. Women should avoid a pregnancy while taking treatment by Lenalidomide or Ibrutinib and for up to 1 month after ending treatment. Men must agree to not to father a child or donate sperm during treatment by Lenalidomide or Ibrutinib and up to 3 months after the last dose of study drug.
10. Women of childbearing potential (WCBP)* must have a negative serum (beta-human chorionic gonadotropin [B-hCG]) or urine pregnancy test at inclusion.
11. Signed informed consent, which could be signed by a person on confidence in case the neurologic status of the patient does not allow him to understand and/or to sign.

Exclusion Criteria:

1. Histology other than DLBCL.
2. Positive HIV serology.
3. Active viral infection with Hepatitis B or C virus.
4. Preexisting immunodeficiency and/or organ transplant recipient.
5. Isolated Central Nervous System (CNS) relapse of systemic Non-Hodgkin's Lymphoma.
6. Prior treatment for PCNSL (except corticosteroids).
7. Isolated primary vitreo-retinal lymphoma.
8. Major surgery, within 4 weeks prior to the first dose of study drug. Stereotactic biopsy and vitrectomy are not considered major surgery.
9. History of stroke or intracranial hemorrhage (except minor post biopsy hemorrhage) within 6 months prior to inclusion.
10. Requires anticoagulation with warfarin or equivalent vitamin K antagonists.
11. Requires treatment with strong CYP3A4 inhibitors.
12. Pregnancy or lactation.
13. Clinically significant cardiovascular disease.
14. Any other active malignancy, except basocellular carcinoma and non-invasive cervix cancer.
15. Inclusion in another experimental anti-cancer drug therapy.
16. No social security affiliation.
17. Persons under legal protection.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2020-10-30 (Actual); Primary Completion 2035-02-02 (Estimated); Study Completion 2035-08-30 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) during the first cycle of treatment for each treatment arm. | 1 month
  Occurrence of a Dose Limiting Toxicity (DLT) during the first cycle of treatment for each treatment arm. The phase Ib is a 3+3 dose escalation design
Complete Response (CR) rate including unconfirmed Complete Response (uCR) at the end of the 4 cycles of induction therapy | 4 months
  The primary endpoint for the phase II part of the study is the Complete Response (CR) rate including unconfirmed CR (CR+uCR) at the end of the 4 cycles of induction therapy. Assessment of response will be based on the International Primary Central Nervous System Lymphoma Collaborative Group (IPCG)

SECONDARY OUTCOMES:
Response rates (CR + uCR) after 2 cycles of induction treatment | 2 months
  Assessment of response will be based on the International Primary Central Nervous System Lymphoma Collaborative Group (IPCG)
Overall response (CR + uCR + Partial Response(PR)), stable disease (SD), and primary refractory patients (PD) after 2 cycles of induction treatment | 2 months
  Assessment of response will be based on the International Primary Central Nervous System Lymphoma Collaborative Group (IPCG)
Overall response (CR + uCR + Partial Response(PR)), stable disease (SD), and primary refractory patients (PD) after 4 cycles of induction treatment | 4 months
  Assessment of response will be based on the International Primary Central Nervous System Lymphoma Collaborative Group (IPCG)
Overall Survival (OS) | 142 months
  Overall Survival (OS) will be calculated from the date of randomization to the date of death, whatever the cause. Patients alive at the date of last contact will be censored at this date.
Progression-Free Survival (PFS) | 142 months
  Progression-Free Survival (PFS) will be calculated from the date of randomization to the date of progression or death (if the patient does not progress). Patients alive without progression at the date of last contact will be censored at this date
The severity of the toxicity of treatment induction or ASCT | 7 months
  Toxicity of treatment induction or ASCT will be graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE 5.0) whenever possible and described by system organ class, preferred term
Patients who will receive ASCT | 7 months
  The percentage of patients who will receive ASCT will be presented

CONTACTS AND LOCATIONS:
Overall Officials: Steven LE GOUILL, PhD, Study Director — Institut Curie
Locations (28):
- France (28):
  - CHU Amiens, Amiens
  - CHU Angers, Angers
  - CH côte Basque, Bayonne
  - CHU Besançon, Besançon
  - Institut Bergonié, Bordeaux
  - CHU Caen, Caen
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - CH Colmar, Colmar
  - CHU Créteil, Créteil
  - CHU Dijon, Dijon
  - CHU Grenoble, Grenoble
  - CHRU Lille, Lille
  - CHU Limoges, Limoges
  - CHU Lyon, Lyon
  - CHU La Timone Marseille, Marseille
  - CHU Nancy, Nancy
  - CHU Nantes, Nantes
  - Centre Lacassagne, Nice
  - CHU Nîmes - Carémeau, Nîmes
  - Institut Curie, Paris
  - Hôpital Cochin, Paris
  - CHU Pitié-Salpêtrière, Paris
  - CHU Poitiers, Poitiers
  - CHU Rennes, Rennes
  - Centre Henri Becquerel, Rouen
  - CHU Strasbourg-Hôpital Hautepierre, Strasbourg
  - IUCT -Oncopole, Toulouse
  - CHU Tours, Tours

IPD SHARING:
Plan to Share IPD: Yes
Sponsor will share de-identified data sets generated under the project will be disseminated in accordance with Institut Curie policies.
Supporting Information: Study Protocol, SAP
Time Frame: Data requests can be submitted starting 9 months after last article publication and will be made accessible for up to 12 months.
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a data sharing agreement (DSA).

REFERENCES:
- [Result] Alcantara M, Chevrier M, Jardin F, Schmitt A, Houillier C, Oberic L, Chinot O, Morschhauser F, Peyrade F, Houot R, Hoang-Xuan K, Ghesquieres H, Soussain C. Phase IB part of LOC-R01, a LOC network non-comparative randomized phase IB/II study testing R-MPV in combination with escalating doses of lenalidomide or ibrutinib for newly diagnosed primary central nervous system lymphoma (PCNSL) patients. J Hematol Oncol. 2024 Sep 19;17(1):86. doi: 10.1186/s13045-024-01606-w. PMID 39300447